CLINICAL TRIAL: NCT02105662
Title: A Phase III Open-Label Clinical Trial to Study the Efficacy and Safety of the Combination Regimen Grazoprevir (GZR) and Elbasvir (EBR) in Treatment-Naïve Subjects With Chronic HCV GT1, GT4, and GT6 Infection Who Are Co-Infected With HIV
Brief Title: An Efficacy and Safety Study of Grazoprevir (MK-5172) + Elbasvir (MK-8742) in the Treatment of Chronic Hepatitis C Virus in Participants Who Are Co-Infected With Human Immunodeficiency Virus:C-EDGE CO-INFXN (MK-5172-061)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5172-061; 2014-000342-30 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Grazoprevir+Elbasvir (Experimental): Participants receive a fixed-dose combination (FDC) of grazoprevir 100 mg plus elbasvir 50 mg once daily for 12 weeks and are followed-up for 24 weeks.
  Interventions: Drug: Grazoprevir 100 mg/Elbasvir 50 mg fixed-dose combination tablets

INTERVENTIONS:
Drug: Grazoprevir 100 mg/Elbasvir 50 mg fixed-dose combination tablets — MK-5172A FDC tablet: MK-5172 (100 mg)/MK-8742 (50 mg)
  Other Names: MK-5172A

SUMMARY:
The purpose of this study is to assess the efficacy and safety of grazoprevir (MK-5172) 100 mg in combination with elbasvir (MK-8742) 50 mg in the treatment of chronic hepatitis C virus (HCV) in participants who are co-infected with human immunodeficiency virus (HIV). The primary hypothesis is that the percentage of participants who receive grazoprevir + elbasvir and achieve Sustained Virologic Response after 12 weeks of therapy (SVR12) will be greater than 70%.

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic HCV genotype (GT) 1, GT4, or GT6 infection with no evidence of non-typeable or mixed GT infection (positive for anti-HCV antibody, HCV RNA, or any of the listed GTs at least 6 months prior to screening must be confirmed by screening lab results)
* Treatment naïve for all anti-HCV treatments
* HIV-1 infection documented by laboratory test
* Currently naïve to treatment with any antiretroviral therapy (ART) and have no plans to initiate ART during this study OR on a HIV ART for at least 8 weeks prior to study entry
* Has not experienced any alteration(s) in HIV therapy within 4 weeks of randomization
* Has at least one viable antiretroviral regimen alternative beyond the current regimen in the event of HIV virologic failure or the development of anti-retroviral drug resistance
* Participants of reproductive potential must agree to remain abstinent from heterosexual activity OR use (or have their partner use) acceptable contraception during heterosexual activity while receiving study drug and for 14 days after last dose of study drug.

Exclusion Criteria:

* Evidence of decompensated liver disease manifested by the presence or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs of symptoms of advanced liver disease
* Co-infected with hepatitis B virus
* History of malignancy <=5 years prior to study start except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or is under evaluation for other active or suspected malignancy
* Taking or planning to take any HIV therapy that includes a ritonavir-boosted or unboosted protease inhibitor, efavirenz or etravirine
* Currently participating or has participated in a study with an investigational compound within 30 days of study start and is not willing to refrain from participating in another study during this study
* Clinically-relevant drug or alcohol abuse within 12 months of study start
* Pregnant, breast feeding, or expecting to conceive or donate eggs from Day 1 of the study throughout treatment and 14 days after the last dose of study medication, or longer if dictated by local regulations
* Organ transplants (including hematopoietic stem cell transplants) other than cornea and hair
* Poor venous access
* History of gastric surgery (e.g., stapling, bypass) or history of malabsorption disorders (e.g., celiac sprue disease)
* Medical condition requiring, or likely to require, chronic systemic administration of corticosteroids during this study
* History of opportunistic infection in the 6 months prior to study start
* Use of HIV drugs other than a dual nucleoside reverse transcriptase inhibitor (NRTI) backbone of tenofovir or abacavir and either emtricitibine or lamivudine PLUS raltegravir (or dolutegravir or rilpivirine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2015-02-20 (Actual); Study Completion 2015-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Rockstroh JK, Nelson M, Katlama C, Lalezari J, Mallolas J, Bloch M, Matthews GV, Saag MS, Zamor PJ, Orkin C, Gress J, Klopfer S, Shaughnessy M, Wahl J, Nguyen BY, Barr E, Platt HL, Robertson MN, Sulkowski M. Efficacy and safety of grazoprevir (MK-5172) and elbasvir (MK-8742) in patients with hepatitis C virus and HIV co-infection (C-EDGE CO-INFECTION): a non-randomised, open-label trial. Lancet HIV. 2015 Aug;2(8):e319-27. doi: 10.1016/S2352-3018(15)00114-9. Epub 2015 Jul 9. PMID 26423374
- [Derived] Asselah T, Reesink H, Gerstoft J, de Ledinghen V, Pockros PJ, Robertson M, Hwang P, Asante-Appiah E, Wahl J, Nguyen BY, Barr E, Talwani R, Serfaty L. Efficacy of elbasvir and grazoprevir in participants with hepatitis C virus genotype 4 infection: A pooled analysis. Liver Int. 2018 Sep;38(9):1583-1591. doi: 10.1111/liv.13727. Epub 2018 Mar 31. PMID 29461687
- [Derived] Reau N, Robertson MN, Feng HP, Caro L, Yeh WW, Nguyen BT, Wahl J, Barr E, Hwang P, Klopfer SO. Concomitant proton pump inhibitor use does not reduce the efficacy of elbasvir/grazoprevir: A pooled analysis of 1,322 patients with hepatitis C infection. Hepatol Commun. 2017 Aug 22;1(8):757-764. doi: 10.1002/hep4.1081. eCollection 2017 Oct. PMID 29404492
- [Derived] Jacobson IM, Lawitz E, Kwo PY, Hezode C, Peng CY, Howe AYM, Hwang P, Wahl J, Robertson M, Barr E, Haber BA. Safety and Efficacy of Elbasvir/Grazoprevir in Patients With Hepatitis C Virus Infection and Compensated Cirrhosis: An Integrated Analysis. Gastroenterology. 2017 May;152(6):1372-1382.e2. doi: 10.1053/j.gastro.2017.01.050. Epub 2017 Feb 11. PMID 28193518

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 218 participants were enrolled and treated on study, 212 participants completed 24 weeks of follow-up.
Groups:
- Grazoprevir+Elbasvir: Participants received a fixed-dose combination (FDC) of grazoprevir 100 mg plus elbasvir 50 mg once daily for 12 weeks and were followed-up for 24 weeks.
Period: Overall Study
Arm/Group | Grazoprevir+Elbasvir
Started | 218
Completed | 212
Not Completed | 6
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Grazoprevir+Elbasvir: Participants received a FDC of grazoprevir 100 mg plus elbasvir 50 mg once daily for 12 weeks and were followed-up for 24 weeks.
Arm/Group | Grazoprevir+Elbasvir
Number analyzed (Participants) | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 183

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks After the End of All Study Therapy (SVR12)
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 (High Pure System). The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a lower limit of quantification of 15 IU/mL and a limit of detection of 9.3 IU/mL (in plasma). SVR12 was defined as undetectable (<9.3 IU/mL) HCV RNA at 12 weeks after the end of all study therapy.
Time Frame: 12 weeks after end of all therapy (Study Week 24)
Population: Full Analysis Set (FAS); all allocated participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Grazoprevir+Elbasvir
Number analyzed (Participants) | 218
percentage of participants | 96.3

2. Primary Outcome: Percentage of Participants Experiencing Adverse Events (AEs) During the Treatment Period and First 14 Follow-up Days
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol -specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Treatment Period plus first 14 follow-up days (up to 14 weeks)
Population: All Participants as Treated (APaT) Population; all participants who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Grazoprevir+Elbasvir
Number analyzed (Participants) | 218
percentage of participants | 73.9

3. Primary Outcome: Percentage of Participants Discontinuing Study Therapy Due to AEs During the Treatment Period
Description: as for outcome 2
Time Frame: Treatment Period (up to 12 weeks)
Population: APaT Population; all participants who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Grazoprevir+Elbasvir
Number analyzed (Participants) | 218
percentage of participants | 0.0

4. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After the End of All Study Therapy (SVR24)
Description: Blood was drawn from each participant to assess HCV RNA plasma levels using the Roche COBAS™ Taqman™ HCV Test, v2.0 (High Pure System). The Roche COBAS Taqman HCV Test, v2.0 assay (High Pure System) had a lower limit of quantification of 15 IU/mL and a limit of detection of 9.3 IU/mL (in plasma). SVR24 was defined as undetectable (<9.3 IU/mL) HCV RNA at 24 weeks after the end of all study therapy.
Time Frame: 24 weeks after end of all therapy (Study Week 36)
Population: FAS; all allocated participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Grazoprevir+Elbasvir
Number analyzed (Participants) | 218
percentage of participants | 93.1

ADVERSE EVENTS:
Time Frame: 12 week treatment period plus 24 week follow-up period (up to 36 weeks)
Description: APaT Population; all participants who received at least one dose of study treatment.
Groups:
- Grazoprevir + Elbasvir: Participants received a FDC of grazoprevir 100 mg plus elbasvir 50 mg once daily for 12 weeks and were followed-up for 24 weeks.
Arm/Group | Grazoprevir + Elbasvir
Serious Adverse Events (participants affected / at risk) | 8/218
Other Adverse Events (participants affected / at risk) | 106/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir + Elbasvir (N=218)
Erysipelas (Infections and infestations) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grazoprevir + Elbasvir (N=218)
Abdominal pain upper (Gastrointestinal disorders) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 18 (19)
Nausea (Gastrointestinal disorders) | 20 (20)
Fatigue (General disorders) | 29 (31)
Nasopharyngitis (Infections and infestations) | 14 (14)
Upper respiratory tract infection (Infections and infestations) | 17 (18)
Headache (Nervous system disorders) | 27 (33)
Insomnia (Psychiatric disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.